CLINICAL TRIAL: NCT00551486
Title: Diagnostic Value of Pyrosequencing for the BRAFV600E Mutation in Ultrasound-Guided Fine-Needle Aspiration Biopsy Samples of Thyroid Incidentalomas
Brief Title: Pyrosequencing of the BRAFV600E Mutation
Status: Completed | Type: Observational
Sponsor: Chungnam National University (Other)
Other Study IDs: 071027
Record Dates: First submitted 2007-10-30; First posted 2007-10-31 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Thyroid Neoplasms
Keywords: Pyrosequencing; BRAFV600E mutation; Thyroid incidentaloma; Ultrasound-guided fine-needle aspiration biopsy
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fine needle aspiration samples of thyroid nodule
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Patients with thyroid incidentaloma underwent ultrasound-guided fine needle aspiration biopsy
  Interventions: Procedure: ultrasound-guided fine needle aspiration biopsy

INTERVENTIONS:
Procedure: ultrasound-guided fine needle aspiration biopsy — Fine needle aspiration (FNA)with cytologic analysis has become a mainstay of thyroid nodule evaluation was used. Nonpalpable nodules were aspirated under ultrasound guidance to facilitate precise targeting of the nodule and to sample the part most likely to improve diagnostic yield.

SUMMARY:
To investigate the diagnostic efficiency of pyrosequencing for the mutant BRAF allele in ultrasound (US)-guided fine needle aspiration biopsies (FNAB) of thyroid incidentalomas.

ELIGIBILITY:
Inclusion Criteria:

* Patients with thyroid nodule larger than 1 cm, or nodule smaller than 1 cm that required further evaluation because of suspicious ultrasound findings

Exclusion Criteria:

* Patients who refuse participation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Patients with thyroid nodule larger than 1 cm, or nodule smaller than 1 cm that required further evaluation because of suspicious ultrasound findings
  2. The average size of the nodules was 1.0 cm.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2006-06; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Minho Shong, M.D., Ph.D., Study Director — Chungnam National University
Locations (1):
- Chungnam National University Hospital, Daejeon, South Korea